CLINICAL TRIAL: NCT05319704
Title: Specificities of the Eccentric Exercise: Energy Expenditure and Nature of Oxidized Substrates
Acronym: Speed-Enso
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RBHP 2018 RICHARD; 2019-A00082-55 (Other: 2019-A00082-55)
Record Dates: First submitted 2021-06-30; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2021-06

CONDITIONS: Overweight; Healthy; Men
Keywords: Energy expenditure; eccentric training; concentric training; oxidized substrates
MeSH Terms: conditions — Overweight; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: participants may receive 4 differents interventions sequentially during the protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test of effort, sub-maximal, progressive, carried out in eccentric mode (Active Comparator): The exercise will start at 10% of VO2max. However, every six minutes, the level of VO2max will be increased by 10%, up to 50%.
  Interventions: Other: Test of effort on cycle on concentric or excentric mode; Other: Kinetics on concentric or excentric mode during test of effort
- Test of effort, sub-maximal, progressive, carried out in concentric mode (Placebo Comparator): The exercise will start at 10% of VO2max. However, every six minutes, the level of VO2max will be increased by 10%, up to 50%.
  Interventions: Other: Test of effort on cycle on concentric or excentric mode; Other: Kinetics on concentric or excentric mode during test of effort
- Kinetic in eccentric mode (Active Comparator): The subjects will have to carry out a test of effort in eccentric or concentric mode during 30 minutes performed at 30% of VO2max.
  The exercise will be followed by indirect oxygen calorimetry (with canopy) extended over a period of 6 hours to measure the energy expenditure, the nature of the oxidized substrates (carbohydrates and lipids) and oxidation rates. During each kinetic, 6 other blood samples will be collected at several times. On these samples, insulin and blood sugar will be measured.
  Interventions: Other: Test of effort on cycle on concentric or excentric mode; Other: Kinetics on concentric or excentric mode during test of effort
- Kinetic in concentric mode (Placebo Comparator): The subjects will have to carry out a test of effort in eccentric or concentric mode during 30 minutes performed at 30% of VO2max.
  The exercise will be followed by indirect oxygen calorimetry (with canopy) extended over a period of 6 hours to measure the energy expenditure, the nature of the oxidized substrates (carbohydrates and lipids) and oxidation rates. During each kinetic, 6 other blood samples will be collected at several times. On these samples, insulin and blood sugar will be measured.
  Interventions: Other: Test of effort on cycle on concentric or excentric mode; Other: Kinetics on concentric or excentric mode during test of effort

INTERVENTIONS:
Other: Test of effort on cycle on concentric or excentric mode — participants may receive 4 interventions sequentially during the protocol
Other: Kinetics on concentric or excentric mode during test of effort — participants may receive 4 interventions sequentially during the protocol

SUMMARY:
Main objective of this clinical trial is to compare the oxidation rates of main carbohydrate and lipid substrates during exercises carried out in eccentric dynamic pedaling mode on a cycloergometer compared to concentric exercises (classic pedaling) at the same oxygen consumption (VO2).

The hypothesis is that lipid oxidation during an eccentric exercise is higher than lipid oxidation during a concentric exercise, done in humans at the capacity of 30% of VO2max.

DETAILED DESCRIPTION:
The written agreement of the subjects will be obtained after information on the aims, nature and possible risks of the study.

Before inclusion, the volunteers will be subjected to a medical check-up at the Nutritional Exploration Unit which includes an examination of personal and family history and current drug treatments, as well as a standard medical examination and a blood test for a biological check-up. Also, the volunteers will be subjected to a check-up with dietetics. Compliance with the inclusion/ exclusion criteria will be verified during this review. Volunteers included in the protocol will go to the Sports Medicine service, or the Nutritional Exploration Unit, or the Clinical Pharmacology Center (CPC) to perform the 11 interventions.

The study will be conducted in 6 periods:

T0 : A standard maximal exercices test performed on an cycloergometer to determine the subject's abilities (VO2) and to set the target powers of the experimental clinical tests. This test will take place in the Sports Medicine service.

T1 : A period of habituation to eccentric exercise, starting from 6 sessions of habituation realized over a period of 15 days where the sessions are gradually increased in duration and intensity. This test will take place in the Sports Medicine service. Before each session of habituation, a Visual Analogue Scale (VAS) will be performed. If the result will be greater than or equal to 3, the session will be rescheduled for another session after 48 hours.

T2 & 3 : Two tests of effort, sub-maximal, progressive, carried out in eccentric mode and concentric mode (each spaced at least 48 hours) to determine the carbohydrate and lipid oxidation rates. Both tests will take place in the Sports Medicine service. The day before each visit, the evening meal will be standardized and eaten before 8 pm. Moreover, the day of both visits, the breakfast will be standardized and eaten 2 hours before the subject will go to Nutritional Exploration Unit.

T4 & 5 : Two exercises tests during 30min performed at 30% VO2max and followed by indirect oxygen calorimetry (with canopy) extended over a period of 6 hours to measure the energy expenditure, the nature of the oxidized substrates (carbohydrates and lipids) and oxidation rates. The day before each visit, the evening meal will be standardized and eaten before 8 pm. Moreover, the day of both visits, the breakfast will be standardized and eaten 2 hours before the subject will go to Nutritional Exploration Unit. In addition, for each kinetic, 7 blood samples will be collected at several times. On these samples, insulin and blood sugar will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers between 20 and 40 years old (20 ≥ years ≤ 40)
* Subjects considered healthy by investigator based on the examination, medical and clinical examination
* Body Mass Index between 27 and 35 kg/m² (27 < BMI < 35)
* Biological check up considered compatible with study participation
* Physical check up considered compatible with study participation (no bones, articular or muscular problems)
* Person who don't smoke and has no treatment
* Person who is in the position to sign informed consent

Exclusion Criteria:

* Smoking
* Person who take any kind of treatments except Paracétamol
* All conditions who have interaction with this clinical trial, or who can deteriorate the exercise capacity or the realization of canopy (claustrophobia)
* Criteria
* Administrative and legal factors
* Person who isn't consent
* Subject not affiliated with social security
* Subject during the exclusion period of a previous study (after verification in the Biomedical Research Volunteers File).

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Measures of oxidation rate of lipid substrates at T2 visit and T3 visit | Through effort test
  The oxidation rate of lipid substrates is measured at 10% of VO2max, 20% of VO2max, 40% of VO2max and 50% of VO2max

SECONDARY OUTCOMES:
Measures of oxidation rate of carbohydrates at T2 visit and T3 visit | Through effort test
  The oxidation rate of carbohydrates is measured at10% of VO2max, 20% of VO2max, 40% of VO2max and 50% of VO2max
Measure of total energy expenditure at T2 visit and T3 visit | Trough exercise
  At the T2 visit and T3 visit, the total energy expenditure is measured
Measure of total energy expenditure at T2 visit and T3 visit | immediatly after exercise
  At the T2 visit and T3 visit, the total energy expenditure is measured
Measure of total energy expenditure at T2 visit and T3 visit | through recovery after exercise, an average of 1 hour
  At the T2 visit and T3 visit, the total energy expenditure is measured
Measure of total energy expenditure | 30 min
  the total energy expenditure is measured during constant-power cycle ergometer tests. This secondary outcome measure will be measured during eccentric and concentric exercises.
Measure of energy expenditure during 6 hours of recovery after exercises | 6 hours
  the energy expenditure is measured during constant-power cycle ergometer tests. This secondary outcome measure will be measured during both kinetics
Measures of substrates oxidation rates at T4 visit and T5 visit | through effort test
  The oxidation rates of substrates are measured during exercises performed at 30% of VO2max
Measures of quantities of oxidized substrates at T4 visit and T5 visit | through effort test
  The quantities of oxidized substrates (carbohydrates, fats, proteins) are measured during exercises
Measures of quantities of carbohydrates at T4 visit and T5 visit | Through energy expenditure measurment an average of 6 hours
  The quantities of oxidized carbohydrates are measured during the measure of energy expenditure
Measures of quantities of fats at T4 visit and T5 visit | Through energy expenditure measurment an average of 6 hours
  The quantities of fats are measured during the measure of energy expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice RANNOU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France